CLINICAL TRIAL: NCT06683586
Title: Brazilian Registry of Chronic Venous Disease - Risk Factors, Comorbidities, Clinical and Surgical Treatment: BRAVO Study
Brief Title: Brazilian Registry of Chronic Venous Disease - Risk Factors, Comorbidities, Clinical and Surgical Treatment
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Vinícius C Quintão, MD, MSc, PhD (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Vinícius C Quintão, MD, MSc, PhD, Assistant Professor, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Other Study IDs: BRAVO
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Venous Disease
Keywords: Chronic Venous Disease; Registry; Venous clinical severity score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: A single group will be included in this cross-sectional study.

SUMMARY:
Chronic venous disease (CVD) is a widespread and challenging condition globally, encompassing the full range of anatomical and functional abnormalities in the venous system of the lower extremities. It is characterized by symptoms such as edema, skin changes, and venous ulcers, primarily caused by venous insufficiency with resulting reflux.

CVD significantly impacts quality of life and imposes a considerable socioeconomic burden. Lifestyle factors play a critical role in the risk of developing CVD. In recent years, average body mass index (BMI) values have risen in Western countries, with obesity recognized as a major risk factor for CVD. Additional factors, including smoking, physical inactivity, and hypertension, are also linked to an increased risk of CVD and chronic venous insufficiency.

There is a lack of recent Brazilian data on the prevalence and epidemiological characteristics of CVD, highlighting the need for this study. This research aims to gather national data on risk factors, associated comorbidities, and treatment types in Brazilian patients with CVD. The primary goal is to describe the clinical and epidemiological profile of CVD in the Brazilian population.

DETAILED DESCRIPTION:
Chronic venous disease (CVD), also known as chronic venous insufficiency in its advanced stages, is marked by dysfunction in the peripheral venous system of the lower extremities, often due to venous flow obstruction or reflux. Affecting approximately 25-45% of women and 10-40% of men, CVD significantly increases public health expenditures. While the exact mechanisms remain unclear, evidence suggests that CVD is multifactorial, involving heightened inflammation, valvular incompetence, and calf muscle dysfunction, all contributing to impaired venous return and elevated venous pressure.

Common symptoms include varicose veins, lower limb edema, leg discomfort, and heaviness. CVD is progressive and can advance from superficial vessel involvement, known as telangiectasia, to deep venous ulcers. Risk factors such as family history, prolonged standing, smoking, and obesity can contribute to its onset and progression. Conservative management focuses on lifestyle changes like exercise, weight control, limb elevation, and compression. Pharmacologic or surgical intervention may be necessary in advanced cases. Left untreated, CVD can severely impact patients' quality of life, hindering daily and work activities.

However, data on CVD prevalence in Brazil is limited, largely based on a single study by Maffei et al. in 1986, which found a 47.6% prevalence of varicose veins and a 3.6% prevalence of advanced CVD in 1,755 adults in Botucatu, São Paulo. To better serve Brazilian patients, further data on CVD prevalence, treatment, and risk factors is essential, aiding healthcare providers in optimizing patient care.

This study aims to characterize the clinical and epidemiological profile of Brazilian CVD patients through a multicenter, prospective observational study. Conducted across 10 centers nationwide, the study will recruit at least 65 patients per center over 12 weeks.

Quality of life will be assessed using the Aberdeen Varicose Vein Questionnaire (AVVQ), with lower scores indicating better quality of life. The Venous Clinical Severity Score (VCSS) will gauge CVD severity, with higher scores indicating greater disease severity. VCSS correlates with the CEAP classification system and ultrasound findings.

CVD diagnoses will be categorized using the CEAP classification:

C0: No signs of venous disease C1: Telangiectasia/reticular veins C2: Varicose veins (≥3 mm diameter) C3: Edema C4: Skin/subcutaneous changes due to CVD, subdivided into C4a (pigmentation/eczema), C4b (lipodermatosclerosis/Atrophie Blanche), and C4c (corona phlebectatica) C5: Healed venous ulcer C6: Active venous ulcer C6r: Recurrent active venous ulcer During exams, patients will undergo physical evaluation for CVD signs, followed by duplex ultrasound of superficial and perforating veins. These will be conducted in both standing and supine positions by qualified vascular specialists, alongside personal medical history, demographics, occupation, physical stress, and varicose vein symptoms.

The study will measure factors including:

Presence and location of saphenous vein insufficiency, reflux, and vein caliber Presence of perforating veins and reflux characteristics Presence of deep vein thrombosis and related complications The study also covers therapeutic procedures such as sclerotherapy, endovenous ablation, and surgical vein removal. Compression stockings and pharmacological treatments (e.g., diosmin + hesperidin, calcium dobesilate, troxerutin) will be documented, including usage frequency and duration.

Data on cardiovascular diseases, comorbidities (e.g., hypertension, diabetes, dyslipidemia), occupation, and family history of CVD will also be collected, providing comprehensive insights into the risk and impact of CVD on the Brazilian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes diagnosed with chronic venous disease;
* Age equal to or greater than 18 years;
* Signature of the informed consent form.

Exclusion Criteria:

* Non-agreement to participate in the study;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) diagnosed with chronic venous disease.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Classification of Venous Disease | Enrollment until Day 1
  Clinical Classification of Venous Disease system CEAP, clinical (C), etiological (E), anatomical (A) and pathological (P) classification as follows:
  C0 = No visible or palpable signs of venous disease; C1 = Telangiectasia or reticular veins; C2 = Varicose veins; distinguishable from reticular veins by a diameter ≥ 3 mm; C3 = Edema;
  C4 = Changes in skin and subcutaneous tissue secondary to CVD, subdivided into:
  C4a = Pigmentation or eczema; C4b = Lipodermatosclerosis or Atrophie Blanche; C4c = Corona phlebectatica; C5 = Cured venous ulcer; C6 = Active venous ulcer; C6r = Recurrent active venous ulcer.

SECONDARY OUTCOMES:
Aberdeen Varicose Vein Questionnaire | Enrollment until 24 hours
  The quality of life assessment will be performed by the Aberdeen Varicose Vein Questionnaire (AVVQ), consisting of 13 questions totaling a score of 0 to 100 points.
Severity of chronic venous disease | Enrollment until 24 hours
  The severity of chronic venous disease will be assessed by the Venous Clinical Severity Score (VCSS), which includes 10 clinical descriptors (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulceration, ulcer size and use of compressive therapy) scored from 0 to 3 (0 = absent; 1= mild; 2= moderate; 3= severe), which can total 30 points.10 VCSS has been shown to have a positive correlation with CEAP and reflux/obstruction assessed by ultrasound.
Proportion of patients receiving treatment | Enrollment until 24 hours
  Proportion of patients with chronic venous disease who receive clinical and/or surgical treatment
Proportion of associated comorbidities | Enrollment until 24 hours
  Proportion of associated comorbidities in patients with chronic venous disease.
Risk factors rate | Enrollment until 24 hours
  Describe the risk factors for the occurrence of chronic venous disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Kikuchi, MD, PhD, Principal Investigator — Santa Casa de Misericordia de Sao Paulo
Locations (1):
- Hospital das Clinicas HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg. 2000 Jun;31(6):1307-12. doi: 10.1067/mva.2000.107094. PMID 10842165
- [Result] Staniszewska A, Tambyraja A, Afolabi E, Bachoo P, Brittenden J. The Aberdeen varicose vein questionnaire, patient factors and referral for treatment. Eur J Vasc Endovasc Surg. 2013 Dec;46(6):715-8. doi: 10.1016/j.ejvs.2013.08.019. Epub 2013 Sep 7. PMID 24119467
- [Result] Maffei FH, Magaldi C, Pinho SZ, Lastoria S, Pinho W, Yoshida WB, Rollo HA. Varicose veins and chronic venous insufficiency in Brazil: prevalence among 1755 inhabitants of a country town. Int J Epidemiol. 1986 Jun;15(2):210-7. doi: 10.1093/ije/15.2.210. PMID 3721683
- [Result] Silva MJ, Louzada ACS, da Silva MFA, Portugal MFC, Teivelis MP, Wolosker N. Epidemiology of 869,220 varicose vein surgeries over 12 years in Brazil: trends, costs and mortality rate. Ann Vasc Surg. 2022 May;82:1-6. doi: 10.1016/j.avsg.2021.11.016. Epub 2021 Dec 20. PMID 34942339
- [Result] Araujo DN, Ribeiro CT, Maciel AC, Bruno SS, Fregonezi GA, Dias FA. Physical exercise for the treatment of non-ulcerated chronic venous insufficiency. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD010637. doi: 10.1002/14651858.CD010637.pub3. PMID 37314059
- [Result] Bradbury A, Evans C, Allan P, Lee A, Ruckley CV, Fowkes FG. What are the symptoms of varicose veins? Edinburgh vein study cross sectional population survey. BMJ. 1999 Feb 6;318(7180):353-6. doi: 10.1136/bmj.318.7180.353. PMID 9933194
- [Result] Nogueira JFL, Teixeira-Viana FC, Barboza-Silva BL, Mendes-Pinto D, Rodrigues-Machado MDG. Advanced Levels of Chronic Venous Insufficiency are Related to an Increased in Arterial Stiffness. Ann Vasc Surg. 2023 Oct;96:365-373. doi: 10.1016/j.avsg.2023.03.013. Epub 2023 Mar 31. PMID 37003361
- [Result] Bergan JJ, Pascarella L, Schmid-Schonbein GW. Pathogenesis of primary chronic venous disease: Insights from animal models of venous hypertension. J Vasc Surg. 2008 Jan;47(1):183-92. doi: 10.1016/j.jvs.2007.09.028. PMID 18178472
- [Result] Silva MFAD, Louzada ACS, Teivelis MP, Leiderman DBD, Portugal MFC, Stabellini N, Amaro Junior E, Wolosker N. Varicose Vein Stripping in 66,577 patients in 11 years in public hospitals in Sao Paulo. Rev Assoc Med Bras (1992). 2022 Nov 25;68(12):1657-1662. doi: 10.1590/1806-9282.20220565. eCollection 2022. PMID 36449789
- [Result] Chaitidis N, Kokkinidis DG, Papadopoulou Z, Kyriazopoulou M, Schizas D, Bakoyiannis C. Treatment of chronic venous disorder: A comprehensive review. Dermatol Ther. 2022 Feb;35(2):e15238. doi: 10.1111/dth.15238. Epub 2021 Dec 13. PMID 34859549